CLINICAL TRIAL: NCT00514475
Title: High-dose Therapy With Autologous Stem Cell Support in First Line Treatment of Mantle Cell Lymphoma- 90Y-Ibritumomab Tiuxetan in Combination With BEAM or BEAC to Improve Outcome for Patients Not in CR After Induction Treatment
Brief Title: Zevalin-BEAM/BEAC With Autologous Stem Cell Support as Consolidation in First Line Treatment of Mantle Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Sponsor-Investigator, Oslo University Hospital, MD PhD, Oslo University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2005-002003-17; NCT00505674 (obsolete NCT alias)
Record Dates: First submitted 2007-08-09; First posted 2007-08-10 (Estimated); Last update posted 2012-05-04 (Estimated); Status verified 2008-05

CONDITIONS: Mantle Cell Lymphoma
Keywords: Mantle cell lymphoma; Zevalin; 90Y-ibritumomab tiuxetan; Radioimmunotherapy; High-dose therapy; First line
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — ibritumomab tiuxetan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: 90Y-ibritumomab tiuxetan (Zevalin) — 90Y-ibritumomab tiuxetan (Zevalin) at 0.4 mCi/kg is administered one week prior to start high-dose chemotherapy (BEAM/BEAC) in patients who have not achieved CR after induction therapy. Predosing with rituximab 250 mg/m2 one weeks prior to radioimmunotherapy and the same day.

SUMMARY:
The purpose of the study is to determine if outcome for patients with mantle cell lymphoma is improved by adding radioimmunotherapy to high-dose regimen before auto-transplant in patients who are not in CR after induction therapy.

DETAILED DESCRIPTION:
Mantle cell lymphoma is considered to have the worst outcome of all non-Hodgkins lymphomas. Since 1997, the Nordic Lymphoma Group has conducted phase II studies in order to improve the results for this lymphoma subtype. The first study included high-dose therapy with autologous stem cell support in the first line of treatment. The results showed the importance of a high quality response to pre-transplant induction treatment, and that CHOP-based regimen alone did not achieve this. Thus, the second trial was designed to improve remissions by including Rituximab and high-dose Ara-C. Results now show that a high rate of molecular remission in the bone marrow was achieved, and the 3-year FFS was improved in comparison to the first study (80% vs 24%). Furthermore, patient who had a molecular relapse (t(11;14) or IgV-gene) were treated with 4 doses of Rituximab and many converted back to be PCR negative.

The present and thus third phase II study aims to improve the high-dose regimen by adding Zevalin radioimmunotherapy in patients who are not in CR prior to transplant. Data from the last trial show that patients not in CR at this point have a worse outcome (3 year FFS of 63%, vs 85% for CR patients). Monitoring for molecular relapse in the bone marrow will be done, and patients who become PCR positive will be treated with Rituximab in order to evaluate the value of this strategy.

ELIGIBILITY:
Inclusion criteria:

1. Age 18 - 65 years.
2. Histologically confirmed (according to the WHO classification) mantle cell lymphoma stage II-IV at time point of diagnosis. The diagnosis has to be confirmed by phenotypic expression of CD5, CD20 and cyclin-D1 and most cases will have t(11;14) translocation.
3. No previous treatment for lymphoma except radiotherapy or one cycle of any regimen and except patients treated in the previous phase II study who can be transferred to NLG-MCL-III before evaluation at week 15.
4. WHO performance status of 0 - 3.
5. Life expectancy of more than 3 months.
6. Written informed consent.

Exclusion Criteria:

1. Severe cardiac disease: cardiac function grade 3-4 (Appendix 1).
2. Impaired liver, renal or other organ function not caused by lymphoma, which will interfere with the treatment.
3. Pregnancy/lactation
4. Men or woman of reproductive potential not agreeing to use acceptable method of birth control during treatment and for six moths after completion of treatment.
5. Known HIV positivity
6. Any other prior malignancy than non-melanoma skin cancer or stage 0 (in situ) cervical carcinoma.
7. Known seropositivity for HCV, HbsAg or other active infection uncontrolled by treatment.
8. Psychiatric illness or condition which could interfere with their ability to understand the requirements of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2005-11; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Time to treatment failure (TTF) for PR/CRu patients receiving Zevalin-BEAM/BEAC | 3 years

SECONDARY OUTCOMES:
Safety | Whole study
TTF for CR patients receiving BEAM/BEAC | 3 year
Overall survival | 5 year
Time to progression | 3 year
Response rates | 6 months
Value of PET | 6 months
Molecular response rates | 6 months
Molecular response and progression-free survival after Rituximab for molecular relapse | 5 years
Microarray gene expression analysis | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Arne Kolstad, MD, Study Chair — Nordic Lymphoma Group; Christian Geisler, MD, Principal Investigator — Nordic Lymphoma Group; Erkki Elonen, MD, Principal Investigator — Nordic Lymphoma Group; Anna Laurell, MD, Principal Investigator — Nordic Lymphoma Group
Locations (1):
- Arne Kolstad, Oslo, Oslo County, Norway

REFERENCES:
- [Derived] Kolstad A, Laurell A, Jerkeman M, Gronbaek K, Elonen E, Raty R, Pedersen LB, Loft A, Bogsrud TV, Kimby E, Hansen PB, Fagerli UM, Nilsson-Ehle H, Lauritzsen GF, Lehmann AK, Sundstrom C, Karjalainen-Lindsberg ML, Ralfkiaer E, Ehinger M, Delabie J, Bentzen H, Schildt J, Kostova-Aherdan K, Frederiksen H, Brown Pde N, Geisler CH; Nordic Lymphoma Group. Nordic MCL3 study: 90Y-ibritumomab-tiuxetan added to BEAM/C in non-CR patients before transplant in mantle cell lymphoma. Blood. 2014 May 8;123(19):2953-9. doi: 10.1182/blood-2013-12-541953. Epub 2014 Mar 20. PMID 24652994
- See also: Web site for the Nordic Lymphoma Group — http://www.nordic-lymphoma.org